CLINICAL TRIAL: NCT03868930
Title: Multisite RCT of STEP-Home: A Transdiagnostic Skill-based Community Reintegration Workshop
Acronym: STEP-Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2907-R
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Post-traumatic Stress Disorder; Traumatic Brain Injury; Substance Related Disorders; Depression; Anxiety Disorders; Suicide; Pain
Keywords: Mental health; Veterans health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic; Substance-Related Disorders; Depression; Anxiety Disorders; Suicide; Pain; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the two group interventions: STEP-Home or Present Centered Group Therapy (PCGT). Each cohort will include a minimum of 8 and a maximum of 20 participants who will be randomized to either STEP-Home (n = 4-10 Veterans) or PCGT (n = 4-10 Veterans). After inclusion and exclusion criteria are verified and a cohort of 8 to 20 is available, randomization into STEP-Home or PCGT occurs and participation in the study begins (i.e., Time 1; T1: Pre), during which the investigators will consent, administer the baseline assessments, randomly assign to the STEP-Home or PCGT arm, and schedule the treatment sessions. All participants will be assessed at the following outcome points: Screening, at randomization (T1), during treatment 4-week skills check (T2), during treatment 8-week skills check (T3), post-intervention (T4), and at 3-months follow up (T5).
Who Masked: Participant
Masking Description: Assessments are all self-report, therefore, blinded assessors are not required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STEP-Home (Experimental): The STEP-Home Arm involves a skills-based intervention focused on Emotional Regulation, Problem Solving, and Attention Training strategies.
  Interventions: Behavioral: STEP-Home
- PCGT (Active Comparator): The Present Center Group Therapy (PCGT) Arm involves a nonspecific, supportive intervention, focused on identifying and discussing current life stressors.
  Interventions: Behavioral: PCGT

INTERVENTIONS:
Behavioral: STEP-Home — This group will meet for 2 hours a week for 12 weeks. The core skills of Emotional Regulation (ER) (45-minutes) and Problem Solving (PS) (45-minutes) are introduced and then integrated throughout all Veteran-specific content modules for practice and repetition for 12 weeks. Attention Training (AT) augments PS and ER core skills and is interspersed throughout group and individual sessions.
  Arms: STEP-Home
Behavioral: PCGT — The PCGT group will also meet for 2 hours a week for 12 weeks. It is a nonspecific and supportive intervention to control for the nonspecific benefits of the group experience (e.g., therapist contact, instillation of hope, expectation of improvement). It will focus on identifying and discussing current life stressors that contribute to reintegration difficulties, psychoeducation, and promotion of wellness and physical health.
  Arms: PCGT

SUMMARY:
In this proposal, the investigators extend their previous SPiRE feasibility and preliminary effectiveness study to examine STEP-Home efficacy in a RCT design. This novel therapy will target the specific needs of a broad range of underserved post-9/11 Veterans. It is designed to foster reintegration by facilitating meaningful improvement in the functional skills most central to community participation: emotional regulation (ER), problem solving (PS), and attention functioning (AT). The skills trained in the STEP-Home workshop are novel in their collective use and have not been systematically applied to a Veteran population prior to the investigators' SPiRE study. STEP-Home will equip Veterans with skills to improve daily function, reduce anger and irritability, and assist reintegration to civilian life through return to work, family, and community, while simultaneously providing psychoeducation to promote future engagement in VA care.

The innovative nature of the STEP-Home intervention is founded in the fact that it is: (a) an adaptation of an established and efficacious intervention, now applied to post-9/11 Veterans; (b) nonstigmatizing (not "therapy" but a "skills workshop" to boost acceptance, adherence and retention); (c) transdiagnostic (open to all post-9/11 Veterans with self-reported reintegration difficulties; Veterans often have multiple mental health diagnoses, but it is not required for enrollment); (d) integrative (focus on the whole person rather than specific and often stigmatizing mental and physical health conditions); (e) comprised of Veteran-specific content to teach participants cognitive behavioral skills needed for successful reintegration (which led to greater acceptability in feasibility study); (f) targets anger and irritability, particularly during interactions with civilians; (g) emphasizes psychoeducation (including other available treatment options for common mental health conditions); and (h) challenges beliefs/barriers to mental health care to increase openness to future treatment and greater mental health treatment utilization. Many Veterans who participated in the development phases of this workshop have gone on to trauma or other focused therapies, or taken on vocational (work/school/volunteer) roles after STEP-Home.

The investigators have demonstrated that the STEP-Home workshop is feasible and results in pre-post change in core skill acquisition that the investigators demonstrated to be directly associated with post-workshop improvement in reintegration status in their SPiRE study. Given the many comorbidities of this cohort, the innovative treatment addresses multiple aspects of mental health, cognitive, and emotional function simultaneously and bolsters reintegration in a short-term group to maximize cost-effectiveness while maintaining quality of care.

DETAILED DESCRIPTION:
Post-9/11 Veterans who served in OEF/OIF face many challenges as they re-enter civilian life after structured military careers. Yet, underutilization and resistance to mental health treatment remains a significant problem. Recent investigations of community reintegration problems among returning Veterans found that half of combat Veterans who use Veterans Administration (VA) services reported difficulty in readjusting to civilian life, including difficulty in social functioning, productivity in work and school settings, community involvement, and self-care domains. High rates of marital, family, and cohabitation discord were reported, with 75% reporting a family conflict in the last week. At least one-third reported divorce, dangerous driving and risky behaviors, increased substance use, and impulsivity and anger control problems since deployment. Almost all Veterans expressed interest in receiving services to help readjust to civilian life, and receiving reintegration services at a VA facility was reported as the preferred way to receive help. Mental health and anger problems are often cited as driving Veterans' difficulties readjusting to civilian life. Anger is becoming more widely recognized for its involvement in the psychological adjustment problems of post-9/11 Veterans. Research has shown that anger directly influences treatment outcome. In fact, history of untreated PTSD and aggression have been demonstrated to be pervasive among post-9/11 Veterans who die by suicide in the months before death. Veterans with probable PTSD report more reintegration and anger problems, and greater interest in services than Veterans without. Reintegration and anger problems continue for years post-combat and may not resolve without intervention.

Research on TBI in post-9/11 Veterans underscores the need for programs that utilize an interdisciplinary approach to reintegration. Programs designed to address challenges of Veterans as they reintegrate in vocational environments, particularly integrative approaches, are greatly needed. The STEP-Home intervention provides such a program. STEP-Home includes focused cognitive and emotional regulation skills training and is informed by the most recent research with returning Veterans and available programs focused on reintegration in VA and military settings (e.g., Battlemind training).

Phase 1: Years 1 and 2 The investigators will initiate the study at the Boston VAMC and develop Standard Operating Procedures for the addition of site 2 in Phase 2.

Phase 2: Years 3 and 4 The investigators will initiate the study at the second site, the Houston VAMC, in Year 3. The investigators will apply in Year 2 for IRB approval to initiate site 2.

Hypotheses & Aims

Primary Aim 1. Examine treatment effects of STEP-Home on primary outcomes relative to Present Centered Group Therapy (PCGT):

Hypothesis 1A. Participants randomized into the STEP-Home intervention will show improvement on reintegration, readjustment, and anger post-intervention (expressed by lower scores; less difficulty).

Military to Civilian Questionnaire (M2CQ), Post-Deployment Readjustment Inventory (PDRI), and State-Trait Anger Expression Inventory (STAXI-2) scores post-intervention (T4) < baseline (T1)

Hypothesis 1B. Participants randomized into STEP-Home will show greater improvement in primary outcomes as compared to PCGT.

Change scores baseline (T1) to post-intervention (T4) STEP-Home > PCGT change scores Post-intervention (T4) primary outcome scores STEP-Home < PCGT primary outcome scores (T4)

Primary Aim 2. Examine maintenance of treatment effects on primary outcomes:

Hypothesis 2: Treatment effects will be maintained at follow up in both groups. Differential treatment effect of STEP-Home over PCGT post-intervention (T4) will be maintained at follow up (T5).

Exploratory Aim 1. Explore treatment effects of STEP-Home on measures of mental health, functional and vocational status and cognitive secondary outcomes targeted indirectly in the workshop.

Exploratory Hypothesis 1. Acquisition of core skills (problem solving, emotional regulation, attention training) will mediate the effect of treatment on primary outcomes post-intervention and at follow up.

The successful completion of the aims proposed has the potential to significantly improve skills to foster civilian reintegration in post-9/11Veterans. Furthermore, the STEP-Home SPiRE feasibility study demonstrated that the workshop also serves as a gateway for Veterans who are hesitant to participate in traditional mental health treatments to promote openness and engagement in additional, critically needed, VA services. Given the high rate of treatment resistance in this cohort, developing acceptable interventions that promote treatment engagement and retention, and open the door to future VA care, is necessary to improve functional status and to reduce long-term healthcare costs of untreated mental health illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Post-9/11 Veterans who report some reintegration, readjustment, or anger difficulty

  * i.e., Veterans who report "some difficulty" (Likert rating) on at least one of the primary measures: M2CQ; PDRI; STAXI-2
* 18-75 years old (to avoid outcomes being affected by aging)
* English-speaking (sessions will be conducted in English)
* Agreeing to participate

  * i.e., completion of ICF/HIPAA

Exclusion Criteria:

* schizophreniform disorder/active psychosis
* bipolar disorder
* active suicidality/homicidality requiring crisis intervention
* other severe psychiatric disorders prohibiting appropriate group participation
* neurological diagnosis prohibiting appropriate group participation (excluding TBI)
* current substance dependence
* current participation in any other form of active behavioral therapy at the time of enrollment

  * e.g., Cognitive Processing Therapy, cognitive rehabilitation for mTBI, or other psychotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine B Fortier, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (2):
- United States (2):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fortier CB, Currao A, Kenna A, Kim S, Beck BM, Katz D, Hursh C, Fonda JR. Online Telehealth Delivery of Group Mental Health Treatment Is Safe, Feasible, and Increases Enrollment and Attendance in Post-9/11 U.S. Veterans. Behav Ther. 2022 May;53(3):469-480. doi: 10.1016/j.beth.2021.11.004. Epub 2021 Nov 25. PMID 35473650
- [Background] Fortier CB, Kenna A, Katz D, Kim S, Hursh C, Beck B, Sablone CA, Currao A, Lebas A, Jorge RE, Fonda JR. STEP-Home transdiagnostic group reintegration workshop to improve mental health outcomes for post-9/11 Veterans: Design, methods, and rationale for a randomized controlled behavioral trial. Contemp Clin Trials. 2024 Jun;141:107536. doi: 10.1016/j.cct.2024.107536. Epub 2024 Apr 16. PMID 38614448

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from VA clinical services, community partners (e.g., schools, Vet Centers, Veteran organizations), advertisements on social media (e.g., Facebook, Instagram), and the Veterans Affairs/Department of Defense Identity Repository.
Pre-assignment Details: 195 (138M/57F) post-9/11 U.S. military Veterans were randomized to either 12 sessions of SH or PCGT. Assessments were conducted at baseline, 12 and 24 weeks. Analyses were based on intention to treat.
Period: Intervention & Post-Treatment Assessment
Arm/Group | STEP-Home | PCGT
Started | 100 (Participants randomized to STEP-Home) | 95 (Participants Randomized to PCGT)
Completed | 53 (Completed treatment) | 57 (Completed treatment)
Not Completed | 47 | 38
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 1 | 4
Not completed — Did not start treatment | 18 | 16
Not completed — Withdrawal by Subject | 25 | 17
Period: Follow-Up Assessment
Arm/Group | STEP-Home | PCGT
Started | 53 | 57
Completed | 44 | 45
Not Completed | 9 | 12
Not completed — Lost to Follow-up | 9 | 12

BASELINE CHARACTERISTICS:
Population: Only participants with available baseline data are included in baseline demographic analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | STEP-Home | PCGT | Total
Number analyzed (Participants) | 93 | 91 | 184
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Participants with available baseline data
  Years | 38.2 (10.3) | 39.8 (10.5) | 39.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 68 | 71 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Categories are not mutually exclusive.
  Participants
    White | 62 | 60 | 122
    Black | 19 | 21 | 40
    Asian | 2 | 1 | 3
    American Indian/Alaskan Native | 4 | 4 | 8
    Other | 15 | 7 | 22
    Hispanic | 23 | 22 | 45
Branch of Service [Count of Participants; unit: Participants] — Population: Participants with available baseline data.
  Participants
    Army | 55 | 43 | 98
    Navy | 10 | 12 | 22
    Air Force | 5 | 9 | 14
    Marines | 11 | 10 | 21
    Coast Guard | 3 | 0 | 3
    Missing Data | 6 | 9 | 15
    Multiple Branches | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Military to Civilian Questionnaire
Description: A 16-item measure of post-deployment community reintegration in post-9/11 Veterans. Higher scores indicate greater reintegration and functional difficulties.
  Min: 0, Max: 64
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: Number of participants analyzed indicates number of enrolled participants that completed survey questions at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 93 | 83
score on a scale
  Baseline | 33.8 (13.2) | 34.7 (11.5)
  Post-Intervention | 25.5 (15.3) | 27.1 (11.2)
  Follow-Up | 24.4 (15.5) | 27.7 (11)
Statistical Analysis 1: Comparison: STEP-Home; Hypothesis 1: Participants randomized into the STEP-Home Intervention will show improvement on reintegration (measured by the Military to Civilian Questionnaire). Hypothesis 2: Treatment effects will be maintained at follow-up for both groups; Test type: Superiority; p < .0001, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the STEP-Home group from Baseline (T1) to Post-Treatment (T2)
Statistical Analysis 2: Comparison: STEP-Home; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the STEP-Home group from Baseline (T1) to Follow-Up (T3)
Statistical Analysis 3: Comparison: PCGT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the Present Centered Group Therapy group from Baseline (T1) to Post-Treatment (T2)
Statistical Analysis 4: Comparison: PCGT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the Present Centered Group Therapy group from Baseline (T1) to Follow-Up (T3)

2. Primary Outcome: Post-deployment Readjustment Inventory (Change)
Description: A 36-item measure of readjustment in post-9/11 Veterans with six subscales (career challenges, social difficulties, intimate relationship problems, health concerns, concerns about deployment, and PTSD symptoms). Min and max scores for all the subscales, and the total score, are below. For all, lower scores are better. Total score is calculated by adding the value of all items in all subscales.
  Career: Min: 5, Max: 25 Health: Min: 5, Max: 25 Intimate Relationship: Min: 5, Max: 25 Social readjustment: Min: 7, Max: 35 Concerns about deployment: Min: 6, Max: 30 PTSD symptoms: Min: 8, Max: 40 TOTAL score: Min: 36, Max: 180
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 91 | 83
score on a scale
  Baseline Total Score | 117.1 (32.6) | 121.0 (26.9)
  Post-Treatment Total Score | 107.8 (35.8) | 116.2 (27.4)
  Follow-Up Total Score | 100.0 (37.9) | 111.1 (27.5)
  Baseline Career Challenges | 15.5 (5.7) | 16.6 (4.5)
  Post-Treatment Career Challenges | 13.9 (5.2) | 15.5 (4.7)
  Follow-Up Career Challenges | 12.8 (5.8) | 14.8 (4.4)
  Baseline Health Concerns | 17.0 (5.7) | 18.0 (4.7)
  Post-Treatment Health Concerns | 15.7 (5.6) | 17.3 (4.9)
  Follow-Up Health Concerns | 14.4 (5.7) | 17.4 (5.0)
  Baseline Intimate Relationship Problems | 15.3 (5.6) | 16.0 (5.1)
  Post-Treatment Intimate Relationship Problems | 14.2 (5.6) | 14.8 (4.6)
  Follow-Up Intimate Relationship Problems | 13.3 (5.6) | 13.8 (4.5)
  Baseline Social Readjustment | 23.5 (7.3) | 24.5 (5.9)
  Post-Treatment Social Readjustment | 22.0 (7.5) | 23.8 (5.9)
  Follow-Up Social Readjustment | 20.8 (8.1) | 21.8 (6.0)
  Baseline Concerns About Deployment | 16.8 (6.2) | 17.5 (5.8)
  Post-Treatment Concerns About Deployment | 15.8 (6.4) | 16.6 (5.3)
  Follow-Up Concerns About Deployment | 14.5 (6.2) | 15.6 (5.5)
  Baseline PTSD Symptoms | 28.3 (8.3) | 30.0 (6.6)
  Post-Treatment PTSD Symptoms | 26.2 (9.0) | 28.1 (6.5)
  Follow-Up PTSD Symptoms | 24.3 (9.4) | 27.7 (6.8)
Statistical Analysis 1: Comparison: STEP-Home; Hypothesis 1: Participants randomized into the STEP-Home Intervention will show improvement on readjustment (measured by the Post Deployment Readjustment Inventory). Hypothesis 2: Treatment effects will be maintained at follow-up for both groups Statistical analysis reported on the total score only; Test type: Superiority; p = 0.0044, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the STEP-Home group from Baseline (T1) to Post-Treatment (T2)
Statistical Analysis 2: Comparison: STEP-Home; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < .0001, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the STEP-Home group from Baseline (T1) to Follow-Up (T3)
Statistical Analysis 3: Comparison: PCGT; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0162, t-test, 2 sided — [p-value comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: PCGT; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0009, t-test, 2 sided — [p-value comment as in outcome 1, analysis 4]

3. Primary Outcome: State-Trait Anger Expression Inventory (STAXI-2) (Change)
Description: A 57-item widely used measure to assess state anger, trait anger, and anger expression with three subscales (state anger, trait anger, and anger expression). Min and max scores for the subscales, and the total score, are below. For all, lower scores are better.
  How I Feel Right Now (State Anger): Min: 10, Max: 40, Calculated by summing 15 items in scale How I Generally Feel (Trait Anger): Min: 10, Max: 40, Calculated by summing 15 items in scale When Angry or Furious (Anger expression index): Min: 24, Max: 96, Calculated by summing anger control scores for each item (12 items) and subtracting that from sum of anger expression scores for each item (12 items)
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 90 | 83
score on a scale
  Baseline State Anger | 25.8 (11.2) | 26.2 (9.2)
  Baseline Trait Anger | 21.9 (6.7) | 21.6 (6.2)
  Baseline Anger Index | 43.1 (14.4) | 42.0 (12.9)
  Post-Treatment State Anger | 22.8 (9.0) | 21.4 (7.3)
  Post-Treatment Trait Anger | 19.9 (7.1) | 20.6 (7.0)
  Post-Treatment Anger Index | 40.2 (13.0) | 41.9 (14.7)
  Follow-Up State Anger | 21.7 (10.0) | 21.9 (7.3)
  Follow-Up Trait Anger | 19.3 (6.1) | 18.5 (6.7)
  Follow-Up Anger Index | 37.7 (12.9) | 39.2 (14.5)
Statistical Analysis 1: Comparison: STEP-Home; Hypothesis 1: Participants randomized into the STEP-Home Intervention will show improvement on anger as measured by the State-Trait Anger Expression Inventory (STAXI). Hypothesis 2: Treatment effects will be maintained at follow-up for both groups; Test type: Superiority; p = 0.0140, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the STEP-Home group from Baseline (T1) to Post-Treatment (T2) Trait Anger
Statistical Analysis 2: Comparison: STEP-Home; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1548, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the STEP-Home group from Baseline (T1) to Post-Treatment (T2) State Anger
Statistical Analysis 3: Comparison: STEP-Home; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0302, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the STEP-Home group from Baseline (T1) to Post-Treatment (T2) Anger Expression Index
Statistical Analysis 4: Comparison: PCGT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0158, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the Present Centered Group Therapy group from Baseline (T1) to Post-Treatment (T2) Trait Anger
Statistical Analysis 5: Comparison: PCGT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0034, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the Present Centered Group Therapy group from Baseline (T1) to Post-Treatment (T2) State Anger
Statistical Analysis 6: Comparison: PCGT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.8776, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the Present Centered Group Therapy group from Baseline (T1) to Post-Treatment (T2) Anger Expression Index
Statistical Analysis 7: Comparison: STEP-Home; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0002, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the STEP-Home group from Baseline (T1) to Follow-Up (T3) Trait Anger
Statistical Analysis 8: Comparison: STEP-Home; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0198, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the STEP-Home group from Baseline (T1) to Follow-Up (T3) State Anger
Statistical Analysis 9: Comparison: STEP-Home; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0013, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the STEP-Home group from Baseline (T1) to Follow-Up (T3) Anger Expression Index
Statistical Analysis 10: Comparison: PCGT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < .0001, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the Present Centered Group Therapy Group from Baseline (T1) to Follow-Up (T3) Trait Anger
Statistical Analysis 11: Comparison: PCGT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .0345, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the Present Centered Group Therapy group from Baseline (T1) to Follow-Up (T3) State Anger
Statistical Analysis 12: Comparison: PCGT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.5918, t-test, 2 sided — P-value indicates significance of T-test (α=0.05) for the Present Centered Group Therapy group from Baseline (T1) to Follow-Up (T3) Anger Expression Index

4. Secondary Outcome: Attention-Related Cognitive Errors Scale (ARCES) (Change)
Description: Measure of everyday performance failures arising from brief failures of sustained attention.
  Min: 12, Max: 60 (lower scores are better)
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 55 | 56
score on a scale
  Baseline | 41.9 (12.4) | 42.7 (9.9)
  Post-Treatment | 38.2 (12.7) | 39.6 (12.9)
  Follow-Up | 37.7 (14.1) | 39.0 (11.7)

5. Secondary Outcome: Problem Solving Inventory (PSI) (Change)
Description: Measure of problem solving confidence, approach-avoidance style, and personal control. Min and max scores for all the subscales, and the total score, are below. For all, lower scores are better. Total score calculated by adding the scores of all items.
  Problem-Solving Confidence: Min: 11, Max: 66 Approach-Avoidance Style: Min: 16, Max: 96 Personal Control: Min: 5, Max: 30 TOTAL score: Min: 32, Max: 192
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 55 | 56
score on a scale
  Baseline Total Score | 100.6 (21.9) | 102.6 (21.7)
  Post-Treatment Total Score | 93.1 (22.0) | 94.1 (26.7)
  Follow-Up Total Score | 94.3 (24.0) | 95.3 (24.2)
  Baseline Problem Solving | 31.7 (8.5) | 31.5 (9.1)
  Post-Treatment Problem Solving | 27.3 (9.0) | 31.5 (9.1)
  Follow-Up Problem Solving | 28.2 (10.6) | 28.8 (9.6)
  Baseline Approach Avoidance | 49.4 (13.4) | 51.8 (13.3)
  Post-Treatment Approach Avoidance | 47.4 (11.2) | 47.6 (15.5)
  Follow-Up Approach Avoidance | 47.2 (11.7) | 47.6 (14.2)
  Baseline Personal Control | 20.3 (5.6) | 21.2 (4.8)
  Post-Treatment Personal Control | 18.4 (4.8) | 18.6 (5.6)
  Follow-Up Personal Control | 19.0 (5.0) | 19.0 (4.4)

6. Secondary Outcome: Difficulties in Emotion Regulation Scale (DERS) (Change)
Description: Measure to assess multiple aspects of emotion dysregulation. Min and max scores for all the subscales, and the total score, are below. For all, lower scores are better.
  Nonacceptance of emotional responses: Min: 6, Max: 30 Difficulty engaging in goal-directed behavior: Min: 6, Max: 25 Impulse control difficulties: Min: 6, Max: 30 Lack of emotional awareness: Min: 6, Max: 30 Limited access to emotion regulation strategies: Min: 8, Max: 40 Lack of emotional clarity: Min: 5, Max: 25 TOTAL score: Min: 36, Max: 180, Total score calculated by adding the scores of all items (reverse scoring awareness items).
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 55 | 56
score on a scale
  Baseline Total Score | 104.2 (26.0) | 106.9 (24.3)
  Post-Treatment Total Score | 90.8 (26.1) | 97.6 (25.8)
  Follow-Up Total Score | 89.2 (30.0) | 94.0 (26.4)
  Baseline Non-Acceptance | 16.1 (7.4) | 18.0 (6.5)
  Post-Treatment Non-Acceptance | 15.0 (6.6) | 16.2 (5.9)
  Follow-Up Non-Acceptance | 14.7 (7.4) | 16.1 (7.4)
  Baseline Goals | 17.4 (4.9) | 17.7 (5.4)
  Post-Treatment Goals | 15.5 (5.6) | 16.6 (5.6)
  Follow-Up Goals | 14.7 (6.1) | 15.9 (5.2)
  Baseline Impulse | 15.3 (5.1) | 15.0 (6.3)
  Post-Treatment Impulse | 13.1 (4.4) | 13.5 (5.7)
  Follow-Up Impulse | 12.2 (5.0) | 12.5 (4.8)
  Baseline Awareness | 17.2 (5.6) | 19.0 (4.9)
  Post-Treatment Awareness | 16.2 (5.8) | 17.8 (5.7)
  Follow-Up Awareness | 16.5 (6.5) | 17.4 (5.6)
  Baseline Strategies | 23.3 (8.4) | 22.6 (7.4)
  Post-Treatment Strategies | 19.0 (8.0) | 20.2 (7.4)
  Follow-Up Strategies | 19.0 (8.5) | 19.5 (7.4)
  Baseline Clarity | 13.7 (4.7) | 14.8 (3.5)
  Post-Treatment Clarity | 12.0 (5.1) | 13.4 (4.0)
  Follow-Up Clarity | 12.1 (4.7) | 13.0 (4.3)

7. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5) (Change)
Description: A 20-item measure of PTSD updated for DSM-5. Min: 0, Max: 80 (lower scores are better)
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 87 | 82
score on a scale
  Baseline | 43.5 (20.1) | 44.9 (17.7)
  Post-Intervention | 36.3 (20.7) | 39.6 (19.4)
  Follow-Up | 34.9 (21.6) | 41.0 (20.6)

8. Secondary Outcome: Depression Anxiety and Stress Scale (DASS-21) (Change)
Description: A 21-item measure of current depression, anxiety, and stress. Each subscale Min: 7, Max: 28 (lower scores are better)
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 86 | 82
score on a scale
  Baseline Anxiety | 15.4 (11.6) | 14.6 (10.0)
  Baseline Depression | 18.7 (12.3) | 19.0 (10.5)
  Baseline Stress | 20.7 (10.9) | 20.9 (9.0)
  Post-Intervention Anxiety | 12.7 (11.2) | 12.8 (9.6)
  Post-Intervention Depression | 16.0 (13.1) | 15.7 (10.6)
  Post-Intervention Stress | 17.1 (11.6) | 18.9 (9.4)
  Follow-Up Anxiety | 11.1 (10.6) | 12.8 (10.2)
  Follow-Up Depression | 12.7 (11.4) | 16.3 (10.0)
  Follow-Up Stress | 15.6 (10.4) | 18.8 (8.8)

9. Secondary Outcome: Neurobehavioral Symptoms Inventory (NSI) (Change)
Description: A 22-item measure of current post-concussive symptoms. Total score Min: 0, Max: 88 (lower scores are better), calculated by adding the scores of all of the subscales.
  Vestibular Min: 0, Max: 12 (3 items) Somatosensory Min: 0, Max: 20 (5 items) Affective Min: 0, Max: 24 (6 items) Cognitive Min: 0, Max: 32 (8 items)
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 87 | 82
score on a scale
  Baseline Total Score | 39.2 (19.7) | 39.0 (16.7)
  Post-Intervention Total Score | 30.5 (19.5) | 35.0 (17.9)
  Follow-Up Total Score | 27.9 (19.1) | 36.3 (17.4)
  Baseline Vestibular | 3.3 (3.2) | 3.3 (2.9)
  Post-Treatment Vestibular | 2.5 (2.6) | 3.3 (2.8)
  Follow-Up Vestibular | 2.7 (2.9) | 4.2 (3.2)
  Baseline Somatic | 8.1 (6.6) | 9.0 (5.5)
  Post-Treatment Somatic | 6.6 (6.1) | 8.4 (5.6)
  Follow-Up Somatic | 7.0 (6.3) | 9.2 (5.7)
  Baseline Cognitive | 9.0 (4.0) | 9.4 (4.2)
  Post-Treatment Cognitive | 7.6 (4.9) | 8.0 (4.8)
  Follow-Up Cognitive | 6.6 (4.2) | 7.7 (4.2)
  Baseline Affective | 14.2 (6.3) | 13.4 (5.3)
  Post-Treatment Affective | 11.5 (6.8) | 12.3 (5.6)
  Follow-Up Affective | 9.4 (6.1) | 12.2 (5.7)

10. Secondary Outcome: World Health Organization Disability Assessment Schedule-2.0 (WHODAS-2.0) (Change)
Description: Measures functional states in six domains (understanding and communicating, getting around, self care, getting along with people, life activities (work/school), and participation in society). Possible raw min and max scores are below. For all subscales and total score, data is presented as a computed score in a range from 0-100. This is calculated by taking the raw score for each subscale and total score, dividing it by number of possible points for the relevant questions, and multiplying it by 100. Lower scores are better.
  Understanding and Communicating: Min: 0, Max: 24 Getting Around: Min: 0, Max: 20 Self Care: Min: 0, Max: 16 Getting Along with People: Min: 0, Max: 20 Life Activities: Min: 0, Max: 16 Work-School: Min: 0, Max: 16 Participation: Min: 0, Max: 32 Total Aggregate: Min: 0, Max: 144
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 86 | 82
score on a scale
  Baseline Total Score | 39.2 (20.7) | 38.3 (18.1)
  Post-Treatment Total Score | 31.6 (22.7) | 33.5 (18.0)
  Follow-Up Total Score | 31.0 (21.6) | 33.7 (19.0)
  Baseline Communicating | 38.4 (22.0) | 41.1 (19.0)
  Post-Treatment Communicating | 35.3 (24.6) | 36.5 (21.6)
  Follow-Up Communicating | 31.3 (22.8) | 36.0 (20.6)
  Baseline Getting Around | 27.6 (26.8) | 24.8 (24.9)
  Post-Treatment Getting Around | 24.8 (24.9) | 26.4 (23.1)
  Follow-Up Getting Around | 24.9 (25.1) | 27.8 (25.0)
  Baseline Self-Care | 18.1 (22.7) | 18.4 (19.9)
  Post-Treatment Self-Care | 14.6 (21.0) | 13.9 (17.7)
  Follow-Up Self-Care | 13.8 (17.6) | 14.7 (18.9)
  Baseline Getting Along | 42.8 (25.5) | 46.7 (21.7)
  Post-Treatment Getting Along | 36.9 (27.8) | 40.4 (19.9)
  Follow-Up Getting Along | 34.4 (27.3) | 41.0 (22.6)
  Baseline Work/Activity | 39.8 (26.2) | 44.2 (24.4)
  Post-Treatment Work/Activity | 34.9 (28.6) | 39.7 (27.8)
  Follow-Up Work/Activity | 34.2 (26.4) | 37.2 (26.8)
  Baseline Participation | 41.4 (26.7) | 42.4 (19.8)
  Post-Treatment Participation | 35.9 (26.6) | 36.4 (21.3)
  Follow-Up Participation | 38.3 (27.3) | 38.0 (21.0)

11. Secondary Outcome: Satisfaction With Life Scale (SWLS) (Change)
Description: A 5-item measure of satisfaction with life. Min: 5, Max: 35 (higher scores are better)
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 83 | 82
score on a scale
  Baseline | 15.1 (7.1) | 15.3 (7.5)
  Post-Treatment | 18.0 (7.6) | 16.6 (7.7)
  Follow-Up | 17.8 (8.9) | 17.7 (7.8)

12. Secondary Outcome: Number of Participants Differing in Activity Engagement Over Time (Change)
Description: Assesses engagement in school, work, and life activities. Participants self reported engagement in each category at each time point. Categories are not mutually exclusive, but rather indicate how many participants endorsed participating in each category at each time point.
  A scale is not used in this measure.
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 84 | 82
Participants
  Baseline Work | 42 | 37
  Baseline School/Training Programs | 18 | 26
  Baseline Volunteer Activities | 15 | 19
  Baseline Veteran-Oriented Programs | 29 | 17
  Baseline Community Activities | 17 | 12
  Baseline Socializing | 50 | 46
  Post-Intervention Work: number analyzed (Participants) | 50 | 53
  Post-Intervention Work | 22 | 20
  Post-Intervention School/Training Programs: number analyzed (Participants) | 50 | 53
  Post-Intervention School/Training Programs | 14 | 19
  Post-Intervention Volunteer Activities: number analyzed (Participants) | 50 | 53
  Post-Intervention Volunteer Activities | 17 | 14
  Post-Intervention Veteran-Oriented Programs: number analyzed (Participants) | 50 | 53
  Post-Intervention Veteran-Oriented Programs | 27 | 20
  Post-Intervention Community Activities: number analyzed (Participants) | 50 | 53
  Post-Intervention Community Activities | 12 | 13
  Post-Intervention Socializing: number analyzed (Participants) | 50 | 53
  Post-Intervention Socializing | 34 | 37
  Follow-Up Work: number analyzed (Participants) | 40 | 43
  Follow-Up Work | 18 | 22
  Follow-Up School/Training Programs: number analyzed (Participants) | 40 | 43
  Follow-Up School/Training Programs | 8 | 16
  Follow-Up Volunteer Activities: number analyzed (Participants) | 40 | 43
  Follow-Up Volunteer Activities | 11 | 11
  Follow-Up Veteran-Oriented Programs: number analyzed (Participants) | 40 | 43
  Follow-Up Veteran-Oriented Programs | 15 | 11
  Follow-Up Community Activities: number analyzed (Participants) | 40 | 43
  Follow-Up Community Activities | 14 | 8
  Follow-Up Socializing: number analyzed (Participants) | 40 | 43
  Follow-Up Socializing | 26 | 25

13. Secondary Outcome: Barriers to Employment Success Inventory (BESI) (Change)
Description: A measure of obstacles to employment in five areas (Personal/Financial, Emotional/Physical, Career Decision-Making and Planning, Job-Seeking Knowledge, and Training/Education). Min and max scores for all the subscales, and the total score, are below. For all, lower scores are better. Only total score analyzed, subscales not reported.
  Personal and Financial: Min: 10, Max: 40 Emotional and Physical: Min: 10, Max: 40 Career Decision-Making and Planning: Min: 10, Max: 40 Job-Seeking Knowledge: Min: 10, Max: 40 Training and Education: Min: 10, Max: 40 TOTAL score: Min: 50, Max: 200
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 84 | 81
score on a scale
  Baseline Total Score | 103.5 (33.9) | 101.8 (32.9)
  Post-Treatment Total Score | 90.7 (33.9) | 96.3 (32.1)
  Follow-Up Total Score | 89.0 (35.9) | 88.3 (32.6)

14. Secondary Outcome: Number of Participants Differing in Average Number of Hours Worked (Change)
Description: Change in average number of hours worked per month over time. Participants self-reported average number of hours worked in the month before STEP-Home (baseline), in each month of the intervention/PCGT (measured at post-treatment), and post-treatment monitoring (follow-up).
  A scale is not used in this measure. Each row indicates the number of participants that worked the indicated number of hours at each time point. Rows are mutually exclusive.
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 94 | 88
Participants
  Baseline <1 hour | 53 | 55
  Baseline 1-10 hours/week | 4 | 4
  Baseline 11-20 hours/week | 3 | 6
  Baseline 21-30 hours/week | 5 | 3
  Baseline 31-40 hours/week | 9 | 10
  Baseline >40 hours/week | 20 | 10
  Post-Intervention <1 hour/week: number analyzed (Participants) | 55 | 57
  Post-Intervention <1 hour/week | 33 | 37
  Post-Intervention 1-10 hours/week: number analyzed (Participants) | 55 | 57
  Post-Intervention 1-10 hours/week | 0 | 3
  Post-Intervention 11-20 hours/week: number analyzed (Participants) | 55 | 57
  Post-Intervention 11-20 hours/week | 0 | 4
  Post-Intervention 21-30 hours/week: number analyzed (Participants) | 55 | 57
  Post-Intervention 21-30 hours/week | 2 | 2
  Post-Intervention 31-40 hours/week: number analyzed (Participants) | 55 | 57
  Post-Intervention 31-40 hours/week | 5 | 6
  Post-Intervention >40 hours/week: number analyzed (Participants) | 55 | 57
  Post-Intervention >40 hours/week | 15 | 5
  Follow-Up <1 hour/week: number analyzed (Participants) | 44 | 45
  Follow-Up <1 hour/week | 26 | 23
  Follow-Up 1-10 hours/week: number analyzed (Participants) | 44 | 45
  Follow-Up 1-10 hours/week | 2 | 2
  Follow-Up 11-20 hours/week: number analyzed (Participants) | 44 | 45
  Follow-Up 11-20 hours/week | 2 | 5
  Follow-Up 21-30 hours/week: number analyzed (Participants) | 44 | 45
  Follow-Up 21-30 hours/week | 0 | 2
  Follow-Up 31-40 hours/week: number analyzed (Participants) | 44 | 45
  Follow-Up 31-40 hours/week | 5 | 8
  Follow-Up >40 hours/week: number analyzed (Participants) | 44 | 45
  Follow-Up >40 hours/week | 9 | 5

15. Secondary Outcome: Frontal Systems Behavior Scale (FrSBe) (Change)
Description: Measures apathy, disinhibition, and executive dysfunction. Min and max possible scores for subscales and total score are below. For all, lower scores are better. Total score calculated by adding the scores of all items. Subscale scores calculated by adding the scores of the items in each subscale.
  Apathy Min: 14, Max: 70 Disinhibition Min: 15, Max: 75 Executive Dysfunction Min: 17, Max: 85 Total Score Min: 46, Max: 230
Time Frame: Baseline, Post 12-Week Treatment, Post Treatment (24 week follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STEP-Home | PCGT
Number analyzed (Participants) | 84 | 80
score on a scale
  Baseline Total Score | 124.8 (25.9) | 124.9 (25.8)
  Post-Treatment Total Score | 111.8 (25.6) | 111.9 (25.0)
  Follow-Up Total Score | 109.2 (23.7) | 110.2 (26.1)
  Baseline Apathy | 41.1 (9.8) | 43.2 (9.4)
  Post-Treatment Apathy | 36.2 (9.8) | 38.3 (10.2)
  Follow-Up Apathy | 35.8 (8.8) | 41.8 (9.3)
  Baseline Disinhibition | 37.6 (10.4) | 37.0 (8.4)
  Post-Treatment Disinhibition | 33.2 (9.6) | 31.8 (9.6)
  Follow-Up Disinhibition | 32.3 (9.6) | 31.1 (10.3)
  Baseline Executive Dysfunction | 45.6 (9.0) | 46.5 (8.1)
  Post-Treatment Executive Dysfunction | 42.4 (8.7) | 41.8 (9.3)
  Follow-Up Executive Dysfunction | 41.1 (7.8) | 41.8 (9.3)

ADVERSE EVENTS:
Time Frame: Baseline, post-intervention (12 weeks), follow-up (24 weeks)
Arm/Group | STEP-Home | PCGT
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/95
Other Adverse Events (participants affected / at risk) | 0/100 | 0/95

LIMITATIONS AND CAVEATS:
The study sample is predominantly male and white, so results should not be generalized to other populations. Treatment outcomes were based on participant self-report. Low follow-up assessment rates were observed due to challenges retaining randomized participants who did not initiate treatment or dropped out of treatment over time, as well as lack of completion of assessments by treatment completers (although completion rates are within expectation for the post-9/11 population of Veterans).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03868930/Prot_SAP_000.pdf